CLINICAL TRIAL: NCT00128245
Title: A 24-week Randomized, Double-blind, Multicenter, Parallel-group, Placebo-controlled Evaluation of the Safety and Efficacy of 0.3% and 1% Pimecrolimus Ophthalmic Suspensions Used Twice Daily in Patients With Moderate to Severe Keratoconjunctivitis Sicca
Brief Title: Safety and Efficacy of Pimecrolimus Ophthalmic Suspension in Patients With Moderate to Severe Keratoconjunctivitis Sicca
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CASM981E2205
Record Dates: First submitted 2005-08-05; First posted 2005-08-09 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2014-01

CONDITIONS: Keratoconjunctivitis Sicca
Keywords: KCS; dry eye; pimecrolimus; Keratoconjunctivitis sicca (dry eye syndrome)
MeSH Terms: conditions — Keratoconjunctivitis Sicca; Dry Eye Syndromes | interventions — pimecrolimus

ARMS (4):
- Pimecrolimus 0.3% (Experimental): ASM981 0.3%
  Interventions: Drug: Pimecrolimus
- Pimecrolimus 1% (Experimental): ASM981 1%
  Interventions: Drug: Pimecrolimus
- Vehicle with carbopol (Placebo Comparator)
  Interventions: Drug: Vehicle
- Vehicle without carbopol (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Pimecrolimus
  Other Names: ASM981
  Arms: Pimecrolimus 0.3%; Pimecrolimus 1%
Drug: Vehicle — Placebo
  Arms: Vehicle with carbopol; Vehicle without carbopol

SUMMARY:
This study evaluates the efficacy and safety of 2 doses of pimecrolimus (0.3% and 1%) ophthalmic suspension in a moderate to severe population of keratoconjunctivitis sicca (KCS, dry eye syndrome) patients.

ELIGIBILITY:
Inclusion Criteria:

* History of artificial tear use
* Moderate to severe signs of dry eye
* Moderate to severe ocular discomfort

Exclusion Criteria:

* Patients with uncontrolled systemic or ocular diseases.
* Have any history of refractive surgery
* Use any topical ocular medications other than those dispensed for the study, during the study

Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440
Dates: Start 2004-09; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
12 week's treatment with 2 concentrations of pimecrolimus (0.3% and 1 %)in one sign and one symptom
change from baseline in fluorescein corneal staining and ocular discomfort(worst symptom,VAS)

SECONDARY OUTCOMES:
24 week's treatment with 2 concentrations of pimecrolimus (0.3% and 1 %)on all signs and symptoms
Global assessment of efficacy and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Gary Foulks, Dr., Principal Investigator — University of Louisville, USA
Locations (1):
- Novartis, East Hanover, New Jersey, United States

REFERENCES:
- See also: Novartis patient recruitment website — http://www.novartisclinicaltrials.com/etrials/DiseaseID69/Dry-Eye-clinical-trials.go